CLINICAL TRIAL: NCT03583567
Title: A Randomized Controlled Study Comparing the Prophylactic Effect of histamine1 and Histamine 2 Receptor Blocker in Prevention Systolic Hypotension After Protamine Administration in Cardiac Patient Having Cardiopulmonary Bypass
Brief Title: Effect of Anti-histamine in Prevention Systolic Hypotension After Protamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Si 2018
Record Dates: First submitted 2018-06-07; First posted 2018-07-11 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Protamine Adverse Reaction
Keywords: protamine; antihistamine
MeSH Terms: interventions — Chlorpheniramine; Ranitidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: normal saline will be used as placebo in control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.9% Normal Saline (Placebo Comparator): Syringe No 1 contain normal saline 1 mL Syringe No 2 contain normal saline 2 mL
  Interventions: Drug: 0.9% Normal Saline
- Chlorpheniramine and ranitidine (Experimental): Syringe No 1 contain chlorpheniramine 10 mg (1 mL) Syringe No 2 contain ranitidine 50 mg (2 mL)
  Interventions: Drug: Chlorpheniramine and ranitidine

INTERVENTIONS:
Drug: Chlorpheniramine and ranitidine — Patient will receive intravenous chlorpheniramine and ranitidine prior to protamine.
  Arms: Chlorpheniramine and ranitidine
Drug: 0.9% Normal Saline — Patient will receive normal saline as placebo.
  Arms: 0.9% Normal Saline

SUMMARY:
Protamine remains the anticoagulant of choice for cardiopulmonary bypass (CPB). The process of protamine neutralization of heparin came with the side effects sometimes; it can be life threatening or fetal reaction. The adverse cardiopulmonary response of protamine has been observed during entire history of clinical cardiac surgery. The true mechanism reaction is difficult to defined and the complexity of the clinical situation The classification of protamine reaction has been divided in to main 3 types (transient systemic hypotension secondary to rapid administration, anaphylactic and anaphylactoid reaction and catastrophic pulmonary vasoconstriction.

The reaction from pharmacologic histamine release is the most common type of reaction. Protamine was believed to induce hypotension by this mechanism, and it was demonstrated to release histamine by degranulation of isolated mast cells From the hypothesis that the systemic hypotension cause by the released of histamine. The investigators will measure the serum tryptase which is the enzyme that released from degranulation of human mast cell. Comparing the serum tryptase level of the patient at baseline, 30 min and 60 min after protamine was given.

There for the hypothesis of this study is administrating of H1 and H2 blocker helps attenuate the drop in MAP after protamine is given.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-3
* Schedule for open heart surgery

Exclusion Criteria:

* History of allergy to the study drugs or protamine
* History of previous cardiac surgery or received protamine
* History of diabetes with insulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 37 minutes
  Systolic and diastolic blood pressure will be recorded every minutes since the start of protamine infusion (in 7 minutes) til 30 minutes after infusion.

SECONDARY OUTCOMES:
Serum tryptase | 60 minutes
  Serum tryptase will be measured before the administration of protamine and at 30 minutes and 60 minutes after protamine

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suksompong S, Wongsripuemtet P, Srinoulprasert Y, Khamtuikrua C, Chaikittisilpa N. H1 and H2 antihistamines pretreatment for attenuation of protamine reactions after cardiopulmonary bypass: a randomized-controlled study. Ann Palliat Med. 2023 Jan;12(1):47-59. doi: 10.21037/apm-22-714. Epub 2022 Dec 16. PMID 36571171